CLINICAL TRIAL: NCT04016896
Title: Efficacy of a Healthy Lifestyle Intervention to Reduce Depression in Older Spousally-bereaved Adults
Brief Title: Depression Prevention in Older Spousally-bereaved Adults
Acronym: WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah T. Stahl, PhD, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19080030; R01MH118270 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Widowed Elders' Lifestyle after Loss (WELL) (Experimental): Digital monitoring of sleep, meals, physical activity (daily); motivational health coaching (weekly); and web-based performance feedback (in real-time) for 12 weeks.
  Interventions: Behavioral: WIdowed Elders' LIfestyle after Loss (WELL)
- Enhanced Usual Care (Active Comparator): Health education, referral to mental health support, and telephone-delivered support (weekly) for 12 weeks.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: WIdowed Elders' LIfestyle after Loss (WELL) — Digital monitoring of sleep, meals, physical activity (daily); motivational health coaching (weekly); and web-based performance feedback (in real-time) for 12 weeks.
  Arms: Widowed Elders' Lifestyle after Loss (WELL)
Other: Enhanced Usual Care — Health education, referral to mental health support, and telephone-delivered support (weekly) for 12 weeks.
  Arms: Enhanced Usual Care

SUMMARY:
Using an indicated prevention approach, investigators propose to enroll 150 spousally-bereaved adults aged 60 years and older in the first 12 months after spousal death who are at high risk for major depression disorder because of subthreshold symptoms of depression. A confirmatory efficacy trial will be conducted in which participants will be randomly assigned to (a) self-monitor sleep, meals, and physical activity for 12 weeks using digital monitoring plus motivational health coaching (WELL; n=75); or (b) enhanced usual care (EUC, usual care plus study assessments, n=75). Objective actigraphic measures of the 24-hour pattern of day and nighttime activity - known as the rest-activity rhythm - will be measured to evaluate circadian rhythms as a mediator of treatment outcomes. Participants will be assessed at baseline, months 1 & 2, post-intervention, and 3, 6,12, 18-months post-intervention. In addition, the investigators will include a subset of participants bereaved by COVID-19 (or suspected as bereaved by COVID-19). Participants in this subset will undergo the same research procedures as the main cohort. Participants in both the main cohort and subset determined to be fully eligible will be randomized into two groups with a total of: enhanced usual care (EUC; n=75) and WELL (WELL; n=75).

DETAILED DESCRIPTION:
The primary aim of this R01 application is to test the efficacy of a new behavioral intervention that targets the timing and regularity of sleep, meals, and physical activity to stabilize circadian rhythms, for reducing symptoms of depression in older acutely-bereaved adults. This trial began at the onset of the SARS-CoV-2/COVID-19 pandemic when grief and loss where ubiquitous and access to mourning services was limited. To test whether this intervention could reduce the severity of associated psychopathological conditions common after spousal death, we added secondary outcomes of anxiety, complicated grief, and posttraumatic stress.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and older;
* spousally (or partner) bereaved up to 12 months (includes bereaved as a result of COVID-19);
* at-risk for major depressive disorder (MDD), based on high-risk markers defined as subthreshold symptoms of depression (Hamilton Depression Rating Scale score of > or = 9), together with absence of current MDD, post-traumatic stress disorder, or persistent complex bereavement disorder

Exclusion Criteria:

* current Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-5) criteria for syndromal mood, psychosis within the last 12 months;
* dementia/cognitive impairment; Telephone Interview Cognitive Screening (TICS) <19;
* acute suicide risk; based on Herbeck et al. protocol for suicide risk management;
* patients taking new psychotropic medications after spousal death to stabilize depression including antidepressants and benzodiazepines >4 days/week for more than two months. Individuals who have been on a stable dose for at least 1 month and agree not to change during participation, unless it is medically necessary, will be included.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sarah t stahl, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC: WPIC- Bellefield Towers, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kazan J, Lyew T, Croswell E, Buysse DJ, Gebara MA, Karp JF, Krafty RT, Rashied AA, Reynolds CF 3rd, Rollman BL, Smagula SF, Stahl ST. A digital health intervention to stabilize the 24-hour rhythm of sleep, meals, and physical activity for reducing depression among older bereaved spouses: Protocol for a randomized controlled trial. Contemp Clin Trials. 2023 Jan;124:107016. doi: 10.1016/j.cct.2022.107016. Epub 2022 Nov 19. PMID 36414207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from university-affiliated research registries, social media, local hospice organizations, grief support groups, and specialty-care medicine at the University of Pittsburgh Medical Center.
Pre-assignment Details: Participants were randomized 1:1 to intervention or control.
Groups:
- Widowed Elders' Lifestyle After Loss (WELL): Behavioral self-monitoring of sleep, meals, and physical activity via digital diaries (daily); motivational health coaching (weekly); and performance feedback on health goals (in real time), for 3 months.
- Enhanced Usual Care: Health education, referral for mental health and grief support, and telephone delivered support (weekly) for 3 months
Period: Overall Study
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
Started | 75 | 76
Completed | 58 | 66
Not Completed | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Widowed Elders' Lifestyle After Loss (WELL): Behavioral self-monitoring of sleep, meals, and physical activity via digital diaries (daily); motivational health coaching (weekly); and performance feedback on health goals (in real time) for 3 months.
- Total: Total of all reporting groups
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported age
  years | 70.3 (6.8) | 70.3 (7.2) | 70.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported sex
  Participants
    Female | 60 | 61 | 121
    Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 6 | 15
    White | 66 | 68 | 134
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Depressive symptoms [Mean (Standard Deviation); unit: score on a scale] — Total score on the Hamilton Rating Scale for Depression. Score range: 0-52 with higher scores indicate greater depression severity.
  score on a scale | 12.6 (12.3) | 3.0 (3.2) | 12.4 (3.0)
Anxiety symptoms [Mean (Standard Deviation); unit: score on a scale] — Total score on the Generalized Anxiety Disorder - 7. Score range = 0-21 with higher scores indicating greater anxiety severity.
  score on a scale | 4.1 (3.5) | 2.9 (2.9) | 3.5 (3.3)
Complicated grief symptoms [Mean (Standard Deviation); unit: score on a scale] — Total score on the Inventory of Complicated Grief. Score range: 0-76 with higher scores indicating greater complicated grief severity.
  score on a scale | 23.4 (11.1) | 21.9 (10.8) | 22.7 (10.9)
Posttraumatic stress symptoms [Mean (Standard Deviation); unit: score on a scale] — Total score on the PTSD Checklist for DSM-5. Score range = 0-80 with higher scores indicating greater PTSD symptom severity
  score on a scale | 15.4 (10.3) | 14.3 (10.6) | 14.8 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depression Symptom Burden at 3 Months
Description: Depression symptoms measured by the clinician administered Hamilton Rating Scale for Depression
Time Frame: baseline vs. 3 months
Population: Of the 75 randomized to intervention, 58 were retained to month 3. Of the 76 randomized to control, 66 were retained to month 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Widowed Elders' Lifestyle After Loss (WELL): Behavioral self-monitoring of sleep, meals, and physical activity via digital diaries (daily); motivational health coaching (weekly); and performance feedback on health goals (in real time).
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
Number analyzed (Participants) | 58 | 66
score on a scale | 5.6 (4.0) | 7.4 (3.9)
Statistical Analysis 1: Comparison: Widowed Elders' Lifestyle After Loss (WELL) vs Enhanced Usual Care; Test type: Superiority; p < .05, ANCOVA; Mean Difference (Final Values) = 3.70

2. Secondary Outcome: Change From Baseline in Anxiety Symptom Burden at 3 Months
Description: Anxiety symptoms measured with the Generalized Anxiety Disorder - 7
Time Frame: baseline vs. 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
Number analyzed (Participants) | 58 | 66
score on a scale | 1.6 (2.5) | 2.1 (2.8)
Statistical Analysis 1: Comparison: Widowed Elders' Lifestyle After Loss (WELL) vs Enhanced Usual Care; Test type: Superiority; p < .05, ANCOVA; Mean Difference (Final Values) = 11.39

3. Secondary Outcome: Change From Baseline in Complicated Grief Symptom Burden at 3 Months
Description: Complicated grief symptoms measured with the Inventory of Complicated Grief
Time Frame: baseline vs. 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
Number analyzed (Participants) | 58 | 66
score on a scale | 16.5 (9.1) | 16.5 (9.7)
Statistical Analysis 1: Comparison: Widowed Elders' Lifestyle After Loss (WELL) vs Enhanced Usual Care; Test type: Superiority; p < .05, ANCOVA; Mean Difference (Final Values) = 2.01

4. Secondary Outcome: Change From Baseline in Posttraumatic Stress Symptom Burden at 3 Months
Description: Posttraumatic stress symptoms measured with the PTSD Checklist for DSM-5
Time Frame: baseline vs. 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
Number analyzed (Participants) | 58 | 66
score on a scale | 9.5 (9.0) | 10.2 (8.3)
Statistical Analysis 1: Comparison: Widowed Elders' Lifestyle After Loss (WELL) vs Enhanced Usual Care; Test type: Superiority; p < .05, ANCOVA; Median Difference (Final Values) = 2.38

ADVERSE EVENTS:
Time Frame: from enrollment until end of intervention, up to 3 months.
Arm/Group | Widowed Elders' Lifestyle After Loss (WELL) | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/75 | 4/76
Other Adverse Events (participants affected / at risk) | 34/75 | 35/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Widowed Elders' Lifestyle After Loss (WELL) (N=75) | Enhanced Usual Care (N=76)
Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory illness (Infections and infestations) | 0 (0) | 1 (1)
Personal injury (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Widowed Elders' Lifestyle After Loss (WELL) (N=75) | Enhanced Usual Care (N=76)
Surgery (Surgical and medical procedures) | 3 (3) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 8 (11) | 10 (14)
Mood/anxiety disorder (Psychiatric disorders) | 6 (7) | 4 (6)
Personal injury (General disorders) | 5 (5) | 6 (6)
Alcohol use disorders (Psychiatric disorders) | 7 (7) | 6 (6)
Arthritis and/or Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 5 (5)
Infections (Infections and infestations) | 5 (5) | 10 (12)
Bladder Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 3 (3) | 4 (4)
Gastrointestinal problems (Gastrointestinal disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)
Cancer (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lupus (Immune system disorders) | 0 (0) | 1 (1)
Cardiovascular problems (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT04016896/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04016896/ICF_000.pdf